CLINICAL TRIAL: NCT07178626
Title: Association of Biomarkers and Gastric Antral Motility Index With Feeding Intolerance in Critically Ill Patients: the BGM-FI Study
Brief Title: Association of Biomarkers and Gastric Antral Motility Index With Feeding Intolerance in Critically Ill Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: BGM-FI
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-08

CONDITIONS: Critically Ill Patients Who Are Not Allowed to Eat Orally But Can Initiate Enteral Nutrition Within 48 Hours of ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients who initiated enteral nutrition early: Critically ill patients who initiated enteral nutrition early
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — This is a prospective observational study and does not involve any intervention measures

SUMMARY:
When the subjects are admitted to the department, the researchers will monitor potential biomarkers of gastrointestinal injury before administering enteral nutrition (a small amount of blood is drawn, serum is separated by centrifugation, and the serum sample is frozen for final centralized biomarker detection), and measure the antral movement index under ultrasound (300ml of warm water is injected into the stomach before measurement, and then the antral movement is observed for 6 minutes) Then, monitor whether the patient has developed feeding intolerance within 7 days of the ICU

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Presence of one or more organ system failures within 24 hours of ICU admission (SOFA score ≥2)
* Expected ICU stay >48 hours
* Inability to take oral nutrition
* No contraindications to enteral nutrition (EN)

Exclusion Criteria:

* Patients who have already received enteral nutrition prior to gastric antral motility measurement or biomarker collection
* Receiving palliative care with expected death within 48 hours
* Pregnancy
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients who can initiate early enteral nutrition
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The subject developed feeding intolerance within 7 days of the ICU | The first to seventh days in the ICU
  The subject developed feeding intolerance (FI) within 7 days of the ICU
  FI is defined as either:
  * intolerance to EN due to any clinical reason (e.g., vomiting (any visible regurgitation of gastric content irrespective of the amount), high gastric residual volume (a single volume exceeds 200 ml), diarrhea (having three or more loose or liquid stools per day with a stool weight greater than 200-250 g/day (or greater than 250 ml/day)), gastrointestinal GI bleeding (any bleeding into the GI tract lumen, confirmed by macroscopic presence of blood in vomited fluids, gastric aspirate or stool), etc.), or
  * FI should be considered present if at least 20 kcal/kg BW/day via enteral route cannot be reached within 72 h of feeding attempt or if enteral feeding has to be stopped for whatever clinical reason.
Pragmatic Definition of Enteral Feeding Intolerance (EFI) - Sensitivity Analysis of the Primary Outcome | From enrollment (ICU admission) through day 7 of enteral nutrition
  This outcome represents a sensitivity analysis for the primary outcome of feeding intolerance.
  EFI is pragmatically defined as a clinician's decision to reduce the prescribed amount of enteral nutrition (EN) specifically because features of gastrointestinal dysfunction appeared during feeding.
  Results from this pragmatic definition will be analyzed to test the robustness of the primary outcome and will be interpreted only as supportive evidence, not as separate primary or secondary outcomes.

SECONDARY OUTCOMES:
28-day mortality | From the 1st to the 28th day after admission to the ICU
  Whether the patient died on the 28th day after being admitted to the ICU
Nutritional adequacy rate on the 7th day | On the seventh day of admission to the ICU
  The probability of achieving 80% of the calorie target (25 kcal/kg/day) in enteral nutrition on the 7th day in the ICU
Length of stay in the ICU | From enrollment to the patient's departure from the ICU (up to 90 days)
  The duration (in days) of the subjects' hospital stay in the ICU
28-day ventilator-free days | From enrollment (ICU admission) through day 28
  The number of days within the first 28 days after enrollment during which the patient was alive and free from invasive mechanical ventilation.
Incidence of Gastric Retention | From enrollment (ICU admission) through day 7 of enteral nutrition
  The occurrence of gastric retention during the first 7 days of enteral nutrition.
  Gastric retention is defined as a single gastric residual volume >200 mL measured by syringe aspiration method.
  The outcome will be recorded as a binary variable (presence or absence).
Incidence of Diarrhea | From enrollment (ICU admission) through day 7 of enteral nutrition
  having three or more loose or liquid stools per day with a stool weight greater than 200-250 g/day (or greater than 250 ml/day

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, China

IPD SHARING:
Plan to Share IPD: No